CLINICAL TRIAL: NCT04822935
Title: Evaluation of Surgical Methods in Terms of Postoperative Pain in Adolescent Idiopathic Scoliosis
Brief Title: Postoperative Pain in Adolescent Idiopathic Scoliosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/1561
Record Dates: First submitted 2021-01-30; First posted 2021-03-30 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Spinal Instrumentation (No Intervention)
- Vertebral Body Tethering (Experimental)
  Interventions: Procedure: Vertebral Body Tethering

INTERVENTIONS:
Procedure: Vertebral Body Tethering — VBT surgery is a surgery performed by thoracotomy in adolescent idiopathic scoliosis patients.
  Arms: Vertebral Body Tethering

SUMMARY:
Scoliosis is a 3-dimensional, structural deformity of the spine. Idiopathic scoliosis is the most common type and it constitutes 75-80% of all scoliosis. Surgical methods are the most effective way to correct the deformity in patients who cannot achieve adequate improvement with supportive therapy. Adolescent idiopathic scoliosis surgeries are among the most invasive surgeries performed on children and adolescents. Large surgical incision and massive tissue damage cause severe postoperative pain. In this study, we aim to compare posterior instrumentation (PE) and vertebral body tethering (VBT) surgeries performed in adolescent idiopathic scoliosis patients in terms of anesthetic management and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA score 1-3 patients
* Adolescent idiopathic scoliosis patients
* Patients who accepted to be included in the study and received written parental consent

Exclusion Criteria:

* Patients with vertebral anomaly due to a secondary reason
* Patients with a diagnosed syndrome
* Patients with a Cobb angle below 40.
* Patients who undergoing reoperation

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Comparison in terms of postoperative pain | 48 hours
  Opioid consumption and VAS (visual analog scale) (0: no pain, 10: the worst pain imaginable) for measurement of postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Irem Basaran, MD, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology
Locations (1):
- Istanbul University Istanbul Medical Faculty, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Canbolat N, Basaran I, Altun D, Akgul T, Buget MI. Postoperative Pain in Adolescent Idiopathic Scoliosis Surgery: A Randomized Controlled Trial. Pain Physician. 2022 Jul;25(4):E589-E596. PMID 35793183